CLINICAL TRIAL: NCT06373341
Title: Rehabilitation of HAND and Arm Function Using a Meta QUEST-based Virtual Reality Game in ICU Patients
Brief Title: Hand and Arm Rehabilitation Using VR
Acronym: HANDQUEST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, Lise Beumeler, Principal Investigator, Frisius Medisch Centrum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL85317.099.23
Record Dates: First submitted 2024-03-11; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Post-Intensive Care Syndrome; ICU Acquired Weakness
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR training (Experimental): The intervention group will participate in training with a VR-exergame for 4 weeks after inclusion. For this training a Meta Quest VR-headset with a game specifically designed for and with ICU patients that was previously pilot tested for feasibility and safety will be used under supervision of a researcher or caregiver until the patient feels ready to practice alone.
  Interventions: Behavioral: VR training for arm and hand rehabilitation
- Standard care (No Intervention): The control group will receive standard care rehabilitation.

INTERVENTIONS:
Behavioral: VR training for arm and hand rehabilitation — The intervention group will participate in training with a VR-exergame for 4 weeks after inclusion. For this training a Meta Quest VR-headset with a game specifically designed for and with ICU patients that was previously pilot tested for feasibility and safety will be used under supervision of a researcher or caregiver until the patient feels ready to practice alone.
  Arms: VR training

SUMMARY:
Patients admitted to the ICU due to critical illness often experience physical, mental, cognitive, or social issues. Research indicates that inadequate physical recovery is associated with lower handgrip strength, and hand function in ICU patients is lower compared to healthy individuals. To address this, a Virtual Reality (VR) exergame was developed to aid rehabilitation. This study aims to investigate the effect of a 4-week VR-exergame intervention on handgrip strength, hand and arm functionality, balance, mobility, and support needs in ICU patients staying for 48 hours or longer. It is a multicenter mixed-methods randomized controlled trial involving adult ICU patients. The intervention involves a 4-week VR-exergame program. Main study parameters include handgrip strength, hand and arm functionality, range of motion, balance, mobility, and support needs. The burden and risks associated with participation are minimal, as VR-based exercises are deemed safe and voluntary. Overall, the study aims to assess the effect of incorporating VR-based rehabilitation into standard care for ICU patients.

DETAILED DESCRIPTION:
Rationale: Patients admitted to the Intensive Care Unit (ICU) due to critical illness may experience new or increased physical, mental, cognitive or social problems. Research from the MCL showed that patients with inadequate physical recovery after one year also have lower handgrip strength at discharge from the ICU and after three months. In addition, a recent study indicated that hand function after ICU admission is lower than in a healthy control group. Early mobilisation focussing on regain of function is therefore essential in ICU patients. Previously, the MCL and 8D Games developed a Virtual Reality exergame that is safe and feasible to use as an addition to standard care mobilisation in the ICU ward. Although the primary goal of the VR-exergame is to provide personalised and fun options in rehabilitation, it may also have additional benefits when it comes to recovery after critical illness. In addition, the VR-exergame may be a feasible option for performing rehabilitation exercises after hospital discharge.

Objective:

Primary:

To investigate the effect of a 4-week VR-exergame intervention on handgrip strength in patients staying in the ICU for 48 hours or longer compared to standard rehabilitation practices.

Secondary:

To investigate the longer term effect of a 4-week VR-exergame intervention on handgrip strength in patients staying in the ICU for 48 hours or longer compared to standard rehabilitation practices at 12 weeks after baseline.

To investigate the effect of a 4-week VR-exergame intervention on hand and arm functionality in patients staying in the ICU for 48 hours or longer compared to standard rehabilitation practices.

To investigate the effect of a 4-week VR-exergame intervention on balance and mobility in patients staying in the ICU for 48 hours or longer compared to standard rehabilitation practices.

To identify support needs of patients staying in the ICU for 48 hours or longer related to the use of a VR-exergame in hospital and in the home situation.

Study design: Multicentre mixed-methods randomised controlled trial.

Study population: Adult ICU patients with a length of stay in ICU of at least 48 hours.

Intervention: 4-week VR-exergame intervention.

Main study parameters/endpoints: Handgrip strength measured by handheld dynamometer, hand and arm functionality by Stroke Upper Limb Capacity Scale and MRC score, hand and wrist range of motion, balance and mobility by Morton Mobility Index and support needs by observational field notes combined with a semi-structured interview.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: VR-based exercises have been used previously in various patient groups, including ICU-patients, and are a safe addition to standard healthcare. Participation with this training is voluntary and an addition to the standard care physical rehabilitation protocol. Patients can stop the exercise at any moment in time, without having to provide an explanation. The exercise activity will be guided and supervised by a trained researcher. Participation in the study measurements and semi-structured interview will require mental effort, but can be conducted in the patients' current living situation to limit burden. Overall, the expected extent of the burden and risks associated with using this healthcare innovation are limited.

ELIGIBILITY:
Inclusion Criteria:

* Length of stay ICU ≥48 hours
* Lives in catchment area of one of the Frisian hospitals
* Understands the Dutch language
* Intact motor skills of at least one upper extremity

Exclusion Criteria:

* Active delirium (CAM-ICU ≥1)
* Severe cognitive dysfunction
* Internal cardiac defibrillator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Handgrip strength | 4 weeks after baseline
  Handgrip strength measured by handheld dynamometer in kg/m2

SECONDARY OUTCOMES:
Handgrip strength | 12 weeks after baseline
  Handgrip strength measured by handheld dynamometer in kg/m2
Arm and hand functionality | 4 and 12 weeks after baseline
  Arm and hand functionality measured by Stroke Upper Limb Capacity Scale (SULCS)
Arm and hand functionality | 4 and 12 weeks after baseline
  Arm and hand functionality measured by Medical Research Council (MRC) score
Arm and hand range of motion | 4 and 12 weeks after baseline
  Range of motion of arm and hand by goniometric measurement
Balance and mobility | 4 and 12 weeks after baseline
  Balance and mobility measured by Morton Mobility Index score
Support need and experience with VR training | at baseline, 4 weeks and 12 weeks
  Qualitative data obtained from participant observations and interviews on support needs and experience with the VR training

CONTACTS AND LOCATIONS:
Overall Officials: Lise Beumeler, PhD, Principal Investigator — Frisius Medisch Centrum
Locations (1):
- Dept of intensive care, Medical Centre Leeuwarden, Leeuwarden, Provincie Friesland, Netherlands

IPD SHARING:
Plan to Share IPD: No